CLINICAL TRIAL: NCT01078558
Title: A Five Year, Post-marketing Observational Study to Follow-up Patients With Rheumatoid Arthritis or Psoriatic Arthritis Who Are Treated With HUMIRA (Adalimumab)
Brief Title: A Belgian Registry of HUMIRA® (Adalimumab) in Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis ( ProAct )
Acronym: ProAct
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Veeda Clinical Research (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: HUM04-28
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2018-11

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis
Keywords: Multicenter study
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with rheumatic disease: Patients suffering from rheumatoid arthritis, psoriatic arthritis or ankylosing spondylitis

SUMMARY:
This is a five year, post-marketing observational study to follow-up patients with rheumatoid arthritis, psoriatic arthritis or ankylosing spondylitis who are treated with HUMIRA (adalimumab).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ongoing HUMIRA (adalimumab) treatment who have been prescribed HUMIRA (adalimumab) within local reimbursement guidelines.
* Patients must be willing to consent to data being collected and provided to Abbott Laboratories.

Exclusion Criteria:

* Contraindications according to the summary of product characteristics.
* Patients who are actually followed in the ReAlise registry (M03-634 NCT00234884).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatologists
Sampling Method: Probability Sample
Enrollment: 5940 (Actual)
Dates: Start 2004-05-13 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5940 participants (2845 with rheumatoid arthritis [RA], 1128 with psoriatic arthritis [PsA], and 1967 with ankylosing spondylitis [AS]) were enrolled. Twenty of these participants were younger than 18 years old (9 RA participants, 1 PsA participant, and 10 AS participants); these participants were not included in any analysis.
Groups:
- Participants With RA: Participants diagnosed with RA in whom Humira® (adalimumab) was prescribed within local reimbursement guidelines.
- Participants With PsA: Participants diagnosed with PsA in whom Humira® (adalimumab) was prescribed within local reimbursement guidelines.
- Participants With AS: Participants diagnosed with AS in whom Humira® (adalimumab) was prescribed within local reimbursement guidelines.
Period: Overall Study
Arm/Group | Participants With RA | Participants With PsA | Participants With AS
Started | 2836 | 1127 | 1957
Oligoarticular PsA | 0 | 197 | 0
Completed | 818 | 372 | 596
Not Completed | 2018 | 755 | 1361

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With RA | Participants With PsA | Participants With AS | Total
Number analyzed (Participants) | 2836 | 1127 | 1957 | 5920
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant in the AS arm had missing data.
  years
    number analyzed (Participants) | 2836 | 1127 | 1956 | 5919
    (all) | 56.64 (12.96) | 49.52 (12.36) | 43.62 (12.47) | 50.98 (13.95)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2004 | 523 | 903 | 3430
  Male | 787 | 591 | 1033 | 2411
  Missing | 45 | 13 | 21 | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Physician's Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — Physician's assessment of disease activity is measured on a visual analogue scale (VAS) from 0 to 100, with the highest values indicating the worst disease activity. Population: Includes all participants with a Baseline assessment.
  units on a scale
    number analyzed (Participants) | 2579 | 1026 | 1741 | 5346
    (all) | 58.47 (22.93) | 54.58 (22.59) | 59.21 (25.32) | 57.96 (23.73)
Tender Joints [Mean (Standard Deviation); unit: tender joints] — A total of 28 joints were assessed for tenderness. Population: Includes all participants with a Baseline assessment.
  tender joints
    number analyzed (Participants) | 2664 | 1046 | 959 | 4669
    (all) | 13.73 (8.90) | 10.47 (8.34) | 2.40 (4.31) | 10.67 (9.16)
Swollen Joints [Mean (Standard Deviation); unit: swollen joints] — A total of 28 joints were assessed for swelling. Population: Includes all participants with a Baseline assessment.
  swollen joints
    number analyzed (Participants) | 2719 | 1049 | 940 | 4708
    (all) | 10.79 (7.18) | 7.46 (5.37) | 1.44 (3.21) | 8.18 (7.17)
Inflammatory Parameter: C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/dL] — Population: Includes all participants with a Baseline assessment.
  mg/dL
    number analyzed (Participants) | 2437 | 937 | 1528 | 4902
    (all) | 3.68 (8.44) | 2.53 (6.90) | 3.24 (19.11) | 3.32 (12.59)
Inflammatory Parameter: Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: mm/hour] — Population: Includes all participants with a Baseline assessment.
  mm/hour
    number analyzed (Participants) | 2320 | 836 | 1257 | 4413
    (all) | 27.58 (21.84) | 18.87 (18.45) | 21.09 (19.23) | 24.08 (20.84)
Health Assessment Questionnaire (HAQ%) [Mean (Standard Deviation); unit: percentage of maximum HAQ score] — The HAQ score measures quality of life in terms of physical function and consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. In the classical HAQ questionnaire, the potential maximum score (60) indicates the most severe disability and the minimum score (0) indicates no disability. The HAQ% is a typical 'Belgian scoring method,' where the actual total score on 60 is converted to a percentage. The HAQ% is performed by all Belgian rheumatologists and is required for obtaining reimbursement. Population: Includes all participants with a Baseline assessment.
  percentage of maximum HAQ score
    number analyzed (Participants) | 2555 | 845 | 69 | 3469
    (all) | 47.80 (19.22) | 41.01 (18.65) | 40.80 (24.57) | 46.00 (19.43)
Disease Activity Score for 28 Joints (DAS28): RA Participants [Mean (Standard Deviation); unit: score on a scale] — The DAS28 score includes 28 tender joint counts, 28 swollen joint counts, CRP/ESR, and participant's global assessment of disease activity. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. Population: Includes all RA participants with a Baseline assessment.
  score on a scale
    number analyzed (Participants) | 383 | 0 | 0 | 383
    (all) | 5.04 (1.21) |  |  | 5.04 (1.21)
DAS28 Category [Count of Participants; unit: Participants] — The DAS28 score includes 28 tender joint counts, 28 swollen joint counts, CRP/ESR, and participant's global assessment of disease activity. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. Population: Includes all RA participants with a Baseline assessment.
  Participants
    < 2.6: number analyzed (Participants) | 383 | 0 | 0 | 383
    < 2.6 | 16 |  |  | 16
    ≥ 2.6 to ≤ 3.2: number analyzed (Participants) | 383 | 0 | 0 | 383
    ≥ 2.6 to ≤ 3.2 | 4 |  |  | 4
    > 3.2: number analyzed (Participants) | 383 | 0 | 0 | 383
    > 3.2 | 363 |  |  | 363
Body Surface Area (BSA) with PsA [Count of Participants; unit: Participants] — Population: Includes all PsA participants with a Baseline assessment.
  Participants
    < 3% of BSA: number analyzed (Participants) | 0 | 783 | 0 | 783
    < 3% of BSA |  | 353 |  | 353
    3% to 10% of BSA: number analyzed (Participants) | 0 | 783 | 0 | 783
    3% to 10% of BSA |  | 211 |  | 211
    11% to 20% of BSA: number analyzed (Participants) | 0 | 783 | 0 | 783
    11% to 20% of BSA |  | 134 |  | 134
    > 20% of BSA: number analyzed (Participants) | 0 | 783 | 0 | 783
    > 20% of BSA |  | 85 |  | 85
Patient's Numerical Rating Scale for Oligarticular PsA Participants [Mean (Standard Deviation); unit: units on a scale] — Participants used a Numerical Rating Scale of 0 to 10 to assess the most important joint, where 0=no disease activity during the previous days and 10=maximal activity during the previous days. Population: Includes all oligoarticular PsA participants with a Baseline assessment.
  units on a scale
    number analyzed (Participants) | 0 | 94 | 0 | 94
    (all) |  | 6.6 (2.0) |  | 6.6 (2.0)
Physician's Numerical Rating Scale for Oligoarticular PsA Participants [Mean (Standard Deviation); unit: units on a scale] — Physicians used a Numerical Rating Scale of 0 to 10 to assess the most important joint, where 0=no disease activity during the previous days and 10=maximal activity during the previous days. Population: Includes all oligoarticular PsA participants with a Baseline assessment by the physican.
  units on a scale
    number analyzed (Participants) | 0 | 95 | 0 | 95
    (all) |  | 6.2 (2.0) |  | 6.2 (2.0)
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) for AS Participants [Mean (Standard Deviation); unit: units on a scale] — BASDAI score measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness, and is calculated using a questionnaire with 6 questions that the participant completes by marking answers on a 10-centimeter visual analog scale with responses that range from 0 (none) to 10 (very severe). The final BASDAI score ranges from 0 to 10 with higher score indicating more severe symptoms. Population: Includes all AS participants with a Baseline assessment.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 1698 | 1698
    (all) |  |  | 6.2 (1.9) | 6.2 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Physician's Assessment of Disease Activity Over Time
Description: Physician's assessment of disease activity is measured on a visual analogue scale (VAS) from 0 to 100, with the highest values indicating the worst disease activity.
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With RA | Participants With PsA | Participants With AS
Number analyzed (Participants) | 1781 | 687 | 1232
units on a scale
  Month 3 | -34.4 (24.7) | -36.2 (24.8) | -40.2 (28.4)
  Month 6: number analyzed (Participants) | 1682 | 645 | 1036
  Month 6 | -38.6 (26.4) | -40.2 (25.6) | -44.5 (28.7)
  Month 12: number analyzed (Participants) | 1453 | 568 | 974
  Month 12 | -40.4 (27.2) | -43.2 (26.6) | -46.6 (28.7)
  Month 24: number analyzed (Participants) | 1178 | 450 | 771
  Month 24 | -42.4 (26.9) | -42.2 (27.2) | -46.6 (28.7)
  Month 60: number analyzed (Participants) | 565 | 243 | 399
  Month 60 | -44.2 (27.3) | -44.8 (29.3) | -50.2 (29.9)

2. Primary Outcome: Change From Baseline in Tender Joints Over Time
Description: A total of 28 joints were assessed for tenderness.
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Participants With RA | Participants With PsA | Participants With AS
Number analyzed (Participants) | 1959 | 755 | 634
tender joints
  Month 3 | -8.5 (8.0) | -6.8 (7.8) | -1.6 (3.5)
  Month 6: number analyzed (Participants) | 1862 | 706 | 533
  Month 6 | -9.4 (8.6) | -7.6 (7.6) | -1.9 (4.6)
  Month 12: number analyzed (Participants) | 1626 | 615 | 499
  Month 12 | -10.2 (8.9) | -8.0 (7.7) | -1.9 (4.1)
  Month 24: number analyzed (Participants) | 1298 | 513 | 377
  Month 24 | -10.4 (8.9) | -7.9 (7.9) | -2.0 (3.9)
  Month 60: number analyzed (Participants) | 637 | 275 | 202
  Month 60 | -11.2 (8.2) | -8.3 (8.7) | -1.9 (3.2)

3. Primary Outcome: Change From Baseline in Swollen Joints Over Time
Description: A total of 28 joints were assessed for swelling.
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Participants With RA | Participants With PsA | Participants With AS
Number analyzed (Participants) | 1982 | 755 | 623
swollen joints
  Month 3 | -7.3 (6.7) | -5.6 (5.7) | -1.3 (3.1)
  Month 6: number analyzed (Participants) | 1890 | 706 | 518
  Month 6 | -8.2 (7.1) | -6.1 (5.2) | -1.4 (3.4)
  Month 12: number analyzed (Participants) | 1654 | 619 | 490
  Month 12 | -8.5 (7.3) | -6.5 (5.4) | -1.3 (2.9)
  Month 24: number analyzed (Participants) | 1328 | 510 | 367
  Month 24 | -9.0 (7.4) | -6.5 (5.8) | -1.4 (2.8)
  Month 60: number analyzed (Participants) | 638 | 275 | 201
  Month 60 | -9.4 (6.7) | -6.8 (6.4) | -1.4 (2.4)

4. Primary Outcome: Inflammatory Parameter: Change From Baseline in CRP Over Time
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants With RA | Participants With PsA | Participants With AS
Number analyzed (Participants) | 1607 | 568 | 838
mg/dL
  Month 3 | -2.1 (8.0) | -1.6 (7.1) | -2.8 (25.1)
  Month 6: number analyzed (Participants) | 1510 | 531 | 707
  Month 6 | -1.9 (6.7) | -1.8 (9.0) | -2.6 (26.1)
  Month 12: number analyzed (Participants) | 1338 | 474 | 677
  Month 12 | -1.9 (7.3) | -1.6 (5.5) | -2.7 (27.5)
  Month 24: number analyzed (Participants) | 1103 | 408 | 580
  Month 24 | -1.9 (7.0) | -1.2 (9.0) | -1.3 (9.3)
  Month 60: number analyzed (Participants) | 545 | 241 | 320
  Month 60 | -1.6 (13.2) | 0.0 (13.8) | -0.7 (4.6)

5. Primary Outcome: Inflammatory Parameter: Change From Baseline in ESR Over Time
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Participants With RA | Participants With PsA | Participants With AS
Number analyzed (Participants) | 1478 | 497 | 670
mm/hour
  Month 3 | -8.3 (18.3) | -7.0 (17.6) | -11.7 (17.8)
  Month 6: number analyzed (Participants) | 1428 | 458 | 582
  Month 6 | -8.1 (18.8) | -8.1 (18.8) | -10.5 (19.2)
  Month 12: number analyzed (Participants) | 1234 | 402 | 536
  Month 12 | -8.4 (19.4) | -8.7 (18.0) | -10.3 (18.5)
  Month 24: number analyzed (Participants) | 1001 | 337 | 468
  Month 24 | -9.2 (20.5) | -6.2 (22.6) | -8.6 (18.8)
  Month 60: number analyzed (Participants) | 468 | 190 | 235
  Month 60 | -8.6 (19.9) | -5.5 (17.4) | -9.8 (19.9)

6. Primary Outcome: Physical Function: Change From Baseline in HAQ% Over Time
Description: The HAQ score measures quality of life in terms of physical function and consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past 7 days using the following responses: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). In the classical HAQ questionnaire, the potential maximum score (60) indicates the most severe disability and the minimum score (0) indicates no disability. The HAQ% is a typical 'Belgian scoring method,' where the actual total score on 60 is converted to a percentage. The HAQ% is performed by all Belgian rheumatologists and is required for obtaining reimbursement.
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage of maximum HAQ score
Arm/Group | Participants With RA | Participants With PsA | Participants With AS
Number analyzed (Participants) | 1580 | 489 | 38
percentage of maximum HAQ score
  Month 3: number analyzed (Participants) | 1580 | 489 | 36
  Month 3 | -19.4 (18.5) | -19.1 (18.8) | -19.6 (19.3)
  Month 6: number analyzed (Participants) | 1568 | 479 | 38
  Month 6 | -22.9 (20.0) | -23.2 (18.7) | -25.8 (21.9)
  Month 12: number analyzed (Participants) | 1279 | 374 | 30
  Month 12 | -22.7 (21.2) | -24.5 (19.3) | -33.4 (22.7)
  Month 24: number analyzed (Participants) | 1064 | 320 | 23
  Month 24 | -24.4 (21.9) | -24.5 (20.9) | -32.3 (20.7)
  Month 60: number analyzed (Participants) | 524 | 165 | 10
  Month 60 | -25.4 (22.0) | -27.1 (21.8) | -34.9 (24.4)

7. Primary Outcome: Change From Baseline in DAS28 Over Time: RA Participants
Description: The DAS28 score includes 28 tender joint counts, 28 swollen joint counts, CRP/ESR, and participant's global assessment of disease activity. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All RA participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With RA
Number analyzed (Participants) | 198
score on a scale
  Month 3 | -1.77 (1.21)
  Month 6: number analyzed (Participants) | 180
  Month 6 | -2.01 (1.55)
  Month 12: number analyzed (Participants) | 179
  Month 12 | -2.38 (1.29)
  Month 24: number analyzed (Participants) | 134
  Month 24 | -2.29 (1.49)
  Month 60: number analyzed (Participants) | 58
  Month 60 | -2.53 (1.44)

8. Primary Outcome: DAS28 Category Over Time: RA Participants
Description: as for outcome 7
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All RA participants with a Baseline and post-baseline assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With RA
Number analyzed (Participants) | 352
Participants
  Month 3 DAS28 < 2.6: number analyzed (Participants) | 274
  Month 3 DAS28 < 2.6 | 106
  Month 3 DAS28 ≥ 2.6 to ≤ 3.2: number analyzed (Participants) | 274
  Month 3 DAS28 ≥ 2.6 to ≤ 3.2 | 50
  Month 3 DAS28 < 3.2: number analyzed (Participants) | 274
  Month 3 DAS28 < 3.2 | 118
  Month 6 DAS28 < 2.6: number analyzed (Participants) | 281
  Month 6 DAS28 < 2.6 | 135
  Month 6 DAS28 ≥ 2.6 to ≤ 3.2: number analyzed (Participants) | 281
  Month 6 DAS28 ≥ 2.6 to ≤ 3.2 | 49
  Month 6 DAS28 < 3.2: number analyzed (Participants) | 281
  Month 6 DAS28 < 3.2 | 97
  Month 12 DAS28 < 2.6: number analyzed (Participants) | 312
  Month 12 DAS28 < 2.6 | 161
  Month 12 DAS28 ≥ 2.6 to ≤ 3.2: number analyzed (Participants) | 312
  Month 12 DAS28 ≥ 2.6 to ≤ 3.2 | 56
  Month 12 DAS28 < 3.2: number analyzed (Participants) | 312
  Month 12 DAS28 < 3.2 | 95
  Month 24 DAS28 < 2.6 | 195
  Month 24 DAS28 ≥ 2.6 to ≤ 3.2 | 60
  Month 24 DAS28 < 3.2 | 97
  Month 60 DAS28 < 2.6: number analyzed (Participants) | 334
  Month 60 DAS28 < 2.6 | 187
  Month 60 DAS28 ≥ 2.6 to ≤ 3.2: number analyzed (Participants) | 334
  Month 60 DAS28 ≥ 2.6 to ≤ 3.2 | 75
  Month 60 DAS28 < 3.2: number analyzed (Participants) | 334
  Month 60 DAS28 < 3.2 | 72

9. Primary Outcome: BSA With PsA Over Time: PsA Participants
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All PsA participants with a Baseline and post-baseline assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With RA
Number analyzed (Participants) | 538
Participants
  Month 3: < 3% of BSA | 398
  Month 3: 3% to 10% of BSA | 97
  Month 3: 11% to 20% of BSA | 32
  Month 3: > 20% of BSA | 11
  Month 6: < 3% of BSA: number analyzed (Participants) | 471
  Month 6: < 3% of BSA | 378
  Month 6: 3% to 10% of BSA: number analyzed (Participants) | 471
  Month 6: 3% to 10% of BSA | 59
  Month 6: 11% to 20% of BSA: number analyzed (Participants) | 471
  Month 6: 11% to 20% of BSA | 24
  Month 6: > 20% of BSA: number analyzed (Participants) | 471
  Month 6: > 20% of BSA | 10
  Month 12: < 3% of BSA: number analyzed (Participants) | 426
  Month 12: < 3% of BSA | 356
  Month 12: 3% to 10% of BSA: number analyzed (Participants) | 426
  Month 12: 3% to 10% of BSA | 41
  Month 12: 11% to 20% of BSA: number analyzed (Participants) | 426
  Month 12: 11% to 20% of BSA | 27
  Month 12: > 20% of BSA: number analyzed (Participants) | 426
  Month 12: > 20% of BSA | 2
  Month 24: < 3% of BSA: number analyzed (Participants) | 352
  Month 24: < 3% of BSA | 298
  Month 24: 3% to 10% of BSA: number analyzed (Participants) | 352
  Month 24: 3% to 10% of BSA | 38
  Month 24: 11% to 20% of BSA: number analyzed (Participants) | 352
  Month 24: 11% to 20% of BSA | 9
  Month 24: > 20% of BSA: number analyzed (Participants) | 352
  Month 24: > 20% of BSA | 7
  Month 60: < 3% of BSA: number analyzed (Participants) | 212
  Month 60: < 3% of BSA | 195
  Month 60: 3% to 10% of BSA: number analyzed (Participants) | 212
  Month 60: 3% to 10% of BSA | 15
  Month 60: 11% to 20% of BSA: number analyzed (Participants) | 212
  Month 60: 11% to 20% of BSA | 1
  Month 60: > 20% of BSA: number analyzed (Participants) | 212
  Month 60: > 20% of BSA | 1

10. Primary Outcome: Change From Baseline in Patient's Numerical Rating Scale Over Time: Oligoarticular PsA Participants
Description: Participants used a Numerical Rating Scale of 0 to 10 to assess the most important joint, where 0=no disease activity during the previous days and 10=maximal activity during the previous days.
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All oligoarticular PsA participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With PsA
Number analyzed (Participants) | 48
units on a scale
  Month 3: number analyzed (Participants) | 45
  Month 3 | -3.4 (2.4)
  Month 6 | -3.8 (2.7)
  Month 12: number analyzed (Participants) | 32
  Month 12 | -2.8 (5.7)
  Month 24: number analyzed (Participants) | 29
  Month 24 | -4.1 (2.8)
  Month 60: number analyzed (Participants) | 10
  Month 60 | -5.3 (2.4)

11. Primary Outcome: Change From Baseline in Physician's Numerical Rating Scale Over Time: Oligoarticular PsA Participants
Description: Physicians used a Numerical Rating Scale of 0 to 10 to assess the most important joint, where 0=no disease activity during the previous days and 10=maximal activity during the previous days.
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All oligoarticular PsA participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With PsA
Number analyzed (Participants) | 47
units on a scale
  Month 3: number analyzed (Participants) | 43
  Month 3 | -3.8 (2.3)
  Month 6 | -4.3 (2.6)
  Month 12: number analyzed (Participants) | 31
  Month 12 | -3.3 (4.5)
  Month 24: number analyzed (Participants) | 27
  Month 24 | -4.0 (2.6)
  Month 60: number analyzed (Participants) | 10
  Month 60 | -5.2 (2.6)

12. Primary Outcome: Change From Baseline in BASDAI Over Time: AS Participants
Description: BASDAI score measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness, and is calculated using a questionnaire with 6 questions that the participant completes by marking answers on a 10-centimeter visual analog scale with responses that range from 0 (none) to 10 (very severe). The final BASDAI score ranges from 0 to 10 with higher score indicating more severe symptoms.
Time Frame: Baseline, Months 3, 6, 12, 24, 60
Population: All oligoarticular PsA participants with a Baseline and post-baseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AS
Number analyzed (Participants) | 1011
score on a scale
  Month 3 | -3.1 (2.4)
  Month 6: number analyzed (Participants) | 821
  Month 6 | -3.2 (2.4)
  Month 12: number analyzed (Participants) | 775
  Month 12 | -3.4 (2.5)
  Month 24: number analyzed (Participants) | 621
  Month 24 | -3.1 (2.5)
  Month 60: number analyzed (Participants) | 323
  Month 60 | -3.3 (2.8)

13. Primary Outcome: Number of Participants With Adverse Events (AEs) Serious AEs (SAEs), and AEs Leading to Study Drug Discontinuation
Description: An AE is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment. An SAE is an AE that results in death, is life-threatening, results in or prolongs hospitalization, results in congenital anomaly, persistent or significant disability/incapacity, spontaneous or elective abortion, or requires intervention to prevent a serious outcome. The protocol required all SAEs to be actively solicited. Non-serious events were not to be actively solicited, and any non-serious AEs were to be collected as spontaneous reports if AbbVie was notified.
Time Frame: up to 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With RA | Participants With PsA | Participants With AS
Number analyzed (Participants) | 2836 | 1127 | 1957
Participants
  Any AE (Includes SAEs) | 976 | 323 | 493
  Any SAE | 560 | 164 | 210
  Any Fatal AE | 41 | 4 | 9
  Any AE Leading to Study Drug Discontinuation | 577 | 171 | 295

ADVERSE EVENTS:
Time Frame: up to Month 60
Description: The protocol required all SAEs to be actively solicited. Non-serious events were not to be actively solicited, and any non-serious AEs were to be collected as spontaneous reports if AbbVie was notified.
Groups:
- All Participants: Participants diagnosed with RA, PsA or AS in whom Humira® (adalimumab) was prescribed within local reimbursement guidelines.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 54/5920
Serious Adverse Events (participants affected / at risk) | 934/5920
Other Adverse Events (participants affected / at risk) | 0/5920
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=5920)
Anaemia (Blood and lymphatic system disorders) | 17 (17)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1)
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 6 (6)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 14 (14)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 3 (4)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1)
Normochromic anaemia (Blood and lymphatic system disorders) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Pseudolymphoma (Blood and lymphatic system disorders) | 1 (1)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 7 (7)
Angina pectoris (Cardiac disorders) | 14 (14)
Angina unstable (Cardiac disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 3 (3)
Aortic valve stenosis (Cardiac disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Arteritis coronary (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 24 (25)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bundle branch block (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 3 (3)
Bundle branch block right (Cardiac disorders) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac asthma (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 4 (4)
Cardiac failure (Cardiac disorders) | 18 (19)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiac fibrillation (Cardiac disorders) | 1 (1)
Cardiac hypertrophy (Cardiac disorders) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 7 (7)
Cardiomyopathy (Cardiac disorders) | 3 (3)
Cardiomyopathy alcoholic (Cardiac disorders) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 2 (2)
Congestive cardiomyopathy (Cardiac disorders) | 5 (5)
Coronary artery dilatation (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 10 (10)
Coronary artery occlusion (Cardiac disorders) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 6 (7)
Cyanosis (Cardiac disorders) | 2 (2)
Diastolic dysfunction (Cardiac disorders) | 2 (2)
Dilatation atrial (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Heart valve incompetence (Cardiac disorders) | 1 (1)
Intracardiac mass (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (4)
Left ventricular dysfunction (Cardiac disorders) | 5 (5)
Left ventricular hypertrophy (Cardiac disorders) | 2 (2)
Mitral valve calcification (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 5 (5)
Mitral valve prolapse (Cardiac disorders) | 1 (1)
Myocardial calcification (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 12 (12)
Myocardial ischaemia (Cardiac disorders) | 4 (4)
Palpitations (Cardiac disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 2 (2)
Pleuropericarditis (Cardiac disorders) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Rheumatic heart disease (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 6 (6)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular flutter (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Dolichocolon (Congenital, familial and genetic disorders) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 2 (2)
Phimosis (Congenital, familial and genetic disorders) | 1 (1)
Thalassaemia (Congenital, familial and genetic disorders) | 1 (1)
Trisomy 18 (Congenital, familial and genetic disorders) | 1 (1)
Truncus arteriosus persistent (Congenital, familial and genetic disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 9 (9)
Acromegaly (Endocrine disorders) | 1 (1)
Addison's disease (Endocrine disorders) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1)
Basedow's disease (Endocrine disorders) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 1 (1)
Goitre (Endocrine disorders) | 3 (3)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 4 (4)
Thyroid cyst (Endocrine disorders) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1)
Altered visual depth perception (Eye disorders) | 1 (1)
Arcus lipoides (Eye disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 5 (5)
Diplopia (Eye disorders) | 1 (1)
Exophthalmos (Eye disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 2 (2)
Eyelids pruritus (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 2 (2)
Visual acuity reduced (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 5 (5)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Abdominal hernia (Gastrointestinal disorders) | 4 (4)
Abdominal mass (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (10)
Abdominal pain lower (Gastrointestinal disorders) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9)
Abdominal symptom (Gastrointestinal disorders) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 2 (2)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 3 (3)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 6 (6)
Colitis ischaemic (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 13 (13)
Crohn's disease (Gastrointestinal disorders) | 8 (8)
Diaphragmatic hernia (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 25 (26)
Diverticular perforation (Gastrointestinal disorders) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 7 (7)
Gastritis (Gastrointestinal disorders) | 6 (6)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal melanosis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (9)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Ileal ulcer (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 8 (8)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 2 (2)
Intestinal polyp (Gastrointestinal disorders) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1)
Intussusception (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 4 (4)
Mouth swelling (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (12)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 9 (9)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal polyp (Gastrointestinal disorders) | 2 (2)
Regurgitation (Gastrointestinal disorders) | 2 (2)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Spigelian hernia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Tongue coated (Gastrointestinal disorders) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Vasculitis gastrointestinal (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 9 (10)
Adverse event (General disorders) | 1 (1)
Asthenia (General disorders) | 20 (21)
Catheter site phlebitis (General disorders) | 1 (1)
Chest discomfort (General disorders) | 6 (6)
Chest pain (General disorders) | 19 (20)
Chills (General disorders) | 10 (10)
Condition aggravated (General disorders) | 1 (1)
Crepitations (General disorders) | 2 (2)
Cyst (General disorders) | 2 (2)
Death (General disorders) | 8 (8)
Discomfort (General disorders) | 1 (1)
Drug effect decreased (General disorders) | 4 (4)
Drug ineffective (General disorders) | 8 (8)
Drug interaction (General disorders) | 1 (1)
Drug intolerance (General disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 28 (28)
Feeling abnormal (General disorders) | 2 (2)
Feeling cold (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Feeling of body temperature change (General disorders) | 1 (1)
Gait disturbance (General disorders) | 4 (5)
General physical health deterioration (General disorders) | 15 (15)
Generalised oedema (General disorders) | 2 (2)
Hernia (General disorders) | 2 (2)
Hyperthermia (General disorders) | 4 (4)
Ill-defined disorder (General disorders) | 5 (5)
Impaired healing (General disorders) | 5 (5)
Inflammation (General disorders) | 16 (16)
Inflammatory pain (General disorders) | 2 (2)
Influenza like illness (General disorders) | 2 (2)
Injection site erythema (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 1 (1)
Injection site reaction (General disorders) | 3 (3)
Injection site urticaria (General disorders) | 1 (1)
Local reaction (General disorders) | 1 (1)
Malaise (General disorders) | 15 (15)
Mass (General disorders) | 2 (2)
Microlithiasis (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 5 (5)
Multiple-drug resistance (General disorders) | 1 (1)
Necrosis (General disorders) | 2 (2)
No adverse event (General disorders) | 3 (3)
Nodule (General disorders) | 1 (1)
Oedema (General disorders) | 5 (5)
Oedema peripheral (General disorders) | 13 (14)
Pain (General disorders) | 12 (12)
Papillitis (General disorders) | 1 (1)
Paradoxical drug reaction (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 4 (4)
Pyrexia (General disorders) | 38 (39)
Sudden death (General disorders) | 2 (2)
Swelling (General disorders) | 1 (1)
Therapy non-responder (General disorders) | 1 (1)
Treatment noncompliance (General disorders) | 2 (2)
Ulcer (General disorders) | 2 (2)
Unevaluable event (General disorders) | 4 (4)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2)
Biliary cyst (Hepatobiliary disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 8 (8)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 17 (17)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 (1)
Fatty liver alcoholic (Hepatobiliary disorders) | 1 (1)
Gallbladder enlargement (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 3 (3)
Hepatic congestion (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 4 (4)
Hepatitis (Hepatobiliary disorders) | 2 (2)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 2 (2)
Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 2 (2)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Allergic oedema (Immune system disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 11 (11)
Immune system disorder (Immune system disorders) | 1 (1)
Immunodeficiency (Immune system disorders) | 2 (2)
Immunosuppression (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Abscess (Infections and infestations) | 2 (2)
Abscess intestinal (Infections and infestations) | 3 (3)
Abscess limb (Infections and infestations) | 4 (4)
Acute sinusitis (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2)
Appendicitis (Infections and infestations) | 3 (3)
Appendicitis perforated (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 12 (12)
Arthritis infective (Infections and infestations) | 1 (1)
Arthritis salmonella (Infections and infestations) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 2 (2)
Bacterial pyelonephritis (Infections and infestations) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 17 (17)
Bronchopulmonary aspergillosis (Infections and infestations) | 2 (2)
Bursitis infective (Infections and infestations) | 3 (3)
Bursitis infective staphylococcal (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 2 (3)
Cellulitis (Infections and infestations) | 4 (4)
Chronic sinusitis (Infections and infestations) | 3 (3)
Clostridial infection (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1)
Cranial nerve infection (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 3 (3)
Cystitis klebsiella (Infections and infestations) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 3 (3)
Device related infection (Infections and infestations) | 4 (4)
Disseminated tuberculosis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 12 (12)
Ear infection (Infections and infestations) | 2 (2)
Empyema (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2)
Enterobacter infection (Infections and infestations) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 19 (19)
Escherichia infection (Infections and infestations) | 3 (3)
Escherichia sepsis (Infections and infestations) | 5 (5)
Escherichia urinary tract infection (Infections and infestations) | 5 (5)
Extradural abscess (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 4 (4)
Gastroenteritis Escherichia coli (Infections and infestations) | 3 (3)
Gastroenteritis salmonella (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
H1N1 influenza (Infections and infestations) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1)
Hepatitis B reactivation (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 8 (8)
Infected skin ulcer (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 16 (16)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 4 (4)
Intervertebral discitis (Infections and infestations) | 2 (2)
Legionella infection (Infections and infestations) | 1 (1)
Leishmaniasis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 10 (10)
Lymph node tuberculosis (Infections and infestations) | 1 (1)
Lymphangitis (Infections and infestations) | 1 (1)
Mastitis (Infections and infestations) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1)
Meningitis herpes (Infections and infestations) | 1 (1)
Meningitis tuberculous (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4)
Necrotising fasciitis (Infections and infestations) | 1 (1)
Nocardiosis (Infections and infestations) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 5 (6)
Ovarian abscess (Infections and infestations) | 1 (1)
Papilloma viral infection (Infections and infestations) | 1 (1)
Pathogen resistance (Infections and infestations) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Pericarditis tuberculous (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 4 (4)
Peritonsillar abscess (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumocystis jirovecii infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 65 (67)
Pneumonia legionella (Infections and infestations) | 4 (4)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 2 (2)
Post procedural pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 4 (4)
Proteus infection (Infections and infestations) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Pseudomonas infection (Infections and infestations) | 3 (3)
Pulmonary sepsis (Infections and infestations) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 3 (3)
Purulent discharge (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 5 (5)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Pyuria (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 6 (7)
Rhinitis (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 12 (12)
Sepsis syndrome (Infections and infestations) | 1 (1)
Septic arthritis staphylococcal (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 12 (12)
Serratia infection (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 11 (11)
Skin infection (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 6 (6)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Superinfection (Infections and infestations) | 1 (1)
Tick-borne viral encephalitis (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 3 (3)
Tooth abscess (Infections and infestations) | 2 (2)
Toxic shock syndrome (Infections and infestations) | 1 (1)
Toxoplasmosis (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 9 (9)
Tuberculosis gastrointestinal (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 22 (24)
Urinary tract infection bacterial (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 3 (3)
Uterine infection (Infections and infestations) | 1 (1)
Vaginal abscess (Infections and infestations) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 6 (6)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 7 (7)
Wound infection staphylococcal (Infections and infestations) | 3 (3)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4)
Cartilage injury (Injury, poisoning and procedural complications) | 2 (2)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Drug dose omission (Injury, poisoning and procedural complications) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 2 (2)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 31 (32)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 4 (4)
Fractured ischium (Injury, poisoning and procedural complications) | 1 (1)
Gastroparesis postoperative (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 9 (9)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 6 (6)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 5 (5)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Kidney rupture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 (4)
Meniscus injury (Injury, poisoning and procedural complications) | 3 (3)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 3 (3)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (3)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3)
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 (4)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 4 (5)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 7 (7)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 4 (4)
Albumin globulin ratio increased (Investigations) | 1 (1)
Alpha 2 globulin increased (Investigations) | 1 (1)
Angiogram peripheral abnormal (Investigations) | 1 (1)
Anti-cyclic citrullinated peptide antibody (Investigations) | 1 (1)
Antibody test abnormal (Investigations) | 1 (1)
Antinuclear antibody positive (Investigations) | 1 (1)
Biopsy breast abnormal (Investigations) | 1 (1)
Biopsy skin abnormal (Investigations) | 1 (3)
Blood calcium increased (Investigations) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Blood culture positive (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood immunoglobulin M increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
Blood phosphorus decreased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 2 (2)
Blood pressure increased (Investigations) | 2 (2)
Blood prolactin increased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 2 (2)
Blood test abnormal (Investigations) | 1 (1)
Blood thyroid stimulating hormone abnormal (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1)
Body temperature decreased (Investigations) | 1 (1)
Breath sounds abnormal (Investigations) | 3 (3)
Bronchoscopy abnormal (Investigations) | 1 (1)
C-reactive protein abnormal (Investigations) | 2 (2)
C-reactive protein increased (Investigations) | 6 (6)
Carcinoembryonic antigen increased (Investigations) | 1 (1)
Cardiac murmur (Investigations) | 3 (3)
Cardiac murmur functional (Investigations) | 1 (1)
Chest X-ray abnormal (Investigations) | 1 (2)
Colonoscopy abnormal (Investigations) | 1 (1)
Computerised tomogram abnormal (Investigations) | 1 (1)
Double stranded DNA antibody positive (Investigations) | 1 (1)
Drug level increased (Investigations) | 1 (1)
Ejection fraction abnormal (Investigations) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram Q wave abnormal (Investigations) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 1 (1)
Electrocardiogram abnormal (Investigations) | 3 (3)
Electrocardiogram repolarisation abnormality (Investigations) | 1 (1)
Epstein-Barr virus antibody positive (Investigations) | 1 (1)
Exercise electrocardiogram abnormal (Investigations) | 1 (1)
Fibrin D dimer increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
General physical condition abnormal (Investigations) | 4 (4)
Haemoglobin decreased (Investigations) | 2 (2)
Heart rate decreased (Investigations) | 1 (1)
Heart rate irregular (Investigations) | 1 (1)
Heart sounds abnormal (Investigations) | 2 (2)
Hepatic enzyme abnormal (Investigations) | 3 (3)
Hepatic enzyme increased (Investigations) | 3 (3)
Immunology test abnormal (Investigations) | 1 (1)
Inflammatory marker increased (Investigations) | 1 (1)
International normalised ratio abnormal (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 2 (2)
Lipids abnormal (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 8 (8)
Liver function test increased (Investigations) | 1 (1)
Lymphocyte count abnormal (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Nuclear magnetic resonance imaging abnormal (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Protein total decreased (Investigations) | 1 (1)
Pulmonary function test decreased (Investigations) | 1 (1)
Pulse abnormal (Investigations) | 1 (1)
Pulse absent (Investigations) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 4 (4)
Rheumatoid factor increased (Investigations) | 1 (1)
Sleep study (Investigations) | 1 (1)
Sputum abnormal (Investigations) | 1 (1)
Synovial fluid analysis (Investigations) | 1 (1)
Total lung capacity abnormal (Investigations) | 1 (1)
Transaminases abnormal (Investigations) | 1 (1)
Transaminases increased (Investigations) | 3 (3)
Troponin increased (Investigations) | 1 (1)
Ultrasound Doppler abnormal (Investigations) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Venous pressure jugular increased (Investigations) | 1 (1)
Vitamin D decreased (Investigations) | 3 (3)
Weight decreased (Investigations) | 19 (19)
Weight increased (Investigations) | 3 (3)
White blood cells urine positive (Investigations) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Cell death (Metabolism and nutrition disorders) | 1 (1)
Central obesity (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 17 (17)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (6)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 (5)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Fluid intake reduced (Metabolism and nutrition disorders) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6)
Hypophagia (Metabolism and nutrition disorders) | 3 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (2)
Hyposideraemia (Metabolism and nutrition disorders) | 1 (1)
Increased insulin requirement (Metabolism and nutrition disorders) | 1 (1)
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 4 (4)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 5 (5)
Polydipsia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 2 (2)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (29)
Arthritis (Musculoskeletal and connective tissue disorders) | 19 (20)
Arthropathy (Musculoskeletal and connective tissue disorders) | 4 (4)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (22)
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 7 (7)
Calcification of muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Chondropathy (Musculoskeletal and connective tissue disorders) | 2 (2)
Eosinophilic fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 16 (19)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 5 (5)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 4 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 20 (21)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint destruction (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 9 (9)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 7 (7)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 8 (8)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Myopathy (Musculoskeletal and connective tissue disorders) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Osteitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 (19)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 4 (5)
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (14)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 5 (5)
Polychondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 7 (7)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 20 (20)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 9 (9)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 5 (5)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Still's disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 8 (8)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 4 (4)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Tendon pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaplastic large cell lymphoma T- and null-cell types recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Angioimmunoblastic T-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Linitis plastica (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1)
Anosognosia (Nervous system disorders) | 1 (1)
Aphasia (Nervous system disorders) | 2 (2)
Apraxia (Nervous system disorders) | 1 (1)
Axonal neuropathy (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 4 (4)
Brain compression (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 5 (5)
Central nervous system lesion (Nervous system disorders) | 1 (1)
Cerebral disorder (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 4 (4)
Cerebral infarction (Nervous system disorders) | 4 (4)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 13 (13)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 5 (5)
Cognitive disorder (Nervous system disorders) | 3 (3)
Coma (Nervous system disorders) | 7 (7)
Complex regional pain syndrome (Nervous system disorders) | 2 (2)
Dementia (Nervous system disorders) | 1 (1)
Demyelination (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7)
Dyskinesia (Nervous system disorders) | 1 (1)
Dysstasia (Nervous system disorders) | 3 (3)
Encephalitis autoimmune (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 4 (4)
Facial paralysis (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 2 (2)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 18 (18)
Hemiparesis (Nervous system disorders) | 5 (5)
Hemiplegia (Nervous system disorders) | 2 (2)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 4 (4)
Hypokinesia (Nervous system disorders) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 2 (2)
Locked-in syndrome (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (3)
Meningoradiculitis (Nervous system disorders) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1)
Micrographia (Nervous system disorders) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 3 (3)
Nerve compression (Nervous system disorders) | 2 (2)
Nervous system disorder (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Neurodegenerative disorder (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 7 (9)
Parkinson's disease (Nervous system disorders) | 2 (2)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 5 (5)
Poor quality sleep (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 2 (2)
Radicular pain (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 10 (10)
Seizure (Nervous system disorders) | 2 (2)
Sensory disturbance (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 3 (3)
Speech disorder (Nervous system disorders) | 2 (2)
Spinal claudication (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 5 (5)
Thalamus haemorrhage (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 8 (8)
Tremor (Nervous system disorders) | 5 (5)
Vasculitis cerebral (Nervous system disorders) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (3)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Device loosening (Product Issues) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 2 (2)
Affect lability (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1)
Bruxism (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 6 (6)
Depression (Psychiatric disorders) | 13 (14)
Depression suicidal (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Dysphoria (Psychiatric disorders) | 1 (1)
Emotional disorder (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 3 (3)
Mood altered (Psychiatric disorders) | 2 (2)
Nervousness (Psychiatric disorders) | 3 (3)
Psychiatric decompensation (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 9 (9)
Anuria (Renal and urinary disorders) | 2 (2)
Bladder disorder (Renal and urinary disorders) | 1 (1)
Bladder irritation (Renal and urinary disorders) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 3 (4)
Cystitis interstitial (Renal and urinary disorders) | 1 (1)
Diabetic end stage renal disease (Renal and urinary disorders) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hypertensive nephropathy (Renal and urinary disorders) | 2 (2)
Incontinence (Renal and urinary disorders) | 2 (2)
Leukocyturia (Renal and urinary disorders) | 1 (1)
Microalbuminuria (Renal and urinary disorders) | 1 (1)
Nephroangiosclerosis (Renal and urinary disorders) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 13 (14)
Nephrotic syndrome (Renal and urinary disorders) | 2 (2)
Nocturia (Renal and urinary disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 4 (4)
Polyuria (Renal and urinary disorders) | 2 (2)
Prerenal failure (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal atrophy (Renal and urinary disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 16 (17)
Renal impairment (Renal and urinary disorders) | 3 (3)
Renal pain (Renal and urinary disorders) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3)
Breast hyperplasia (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 3 (3)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 2 (2)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 4 (4)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1)
Pelvic haemorrhage (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 2 (2)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (18)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (41)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Rales (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Yawning (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acanthosis (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7)
Excessive skin (Skin and subcutaneous tissue disorders) | 1 (1)
Generalised erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 2 (2)
Hidradenitis (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (6)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Parakeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 11 (11)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin dystrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 (6)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1)
Alcoholic (Social circumstances) | 1 (1)
Bedridden (Social circumstances) | 2 (2)
Impaired driving ability (Social circumstances) | 1 (1)
Impaired work ability (Social circumstances) | 2 (2)
Loss of personal independence in daily activities (Social circumstances) | 3 (3)
Poor personal hygiene (Social circumstances) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1)
Angioplasty (Surgical and medical procedures) | 1 (1)
Arterial catheterisation (Surgical and medical procedures) | 1 (1)
Arterial stent insertion (Surgical and medical procedures) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 6 (6)
Bladder operation (Surgical and medical procedures) | 1 (1)
Bone debridement (Surgical and medical procedures) | 1 (1)
Breast prosthesis removal (Surgical and medical procedures) | 1 (1)
Bunion operation (Surgical and medical procedures) | 1 (1)
Caesarean section (Surgical and medical procedures) | 1 (1)
Cataract operation (Surgical and medical procedures) | 2 (2)
Cholecystectomy (Surgical and medical procedures) | 2 (2)
Corneal transplant (Surgical and medical procedures) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 2 (2)
Coronary artery bypass (Surgical and medical procedures) | 5 (5)
Debridement (Surgical and medical procedures) | 1 (1)
Elbow operation (Surgical and medical procedures) | 1 (1)
Foot operation (Surgical and medical procedures) | 3 (4)
Gastrectomy (Surgical and medical procedures) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 2 (2)
Hip arthroplasty (Surgical and medical procedures) | 26 (26)
Hospitalisation (Surgical and medical procedures) | 10 (10)
Hysterectomy (Surgical and medical procedures) | 2 (2)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 3 (3)
Joint stabilisation (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 22 (23)
Knee operation (Surgical and medical procedures) | 1 (1)
Mammoplasty (Surgical and medical procedures) | 1 (1)
Mastectomy (Surgical and medical procedures) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1)
Meniscus removal (Surgical and medical procedures) | 3 (3)
Metabolic surgery (Surgical and medical procedures) | 1 (1)
Metatarsal excision (Surgical and medical procedures) | 1 (1)
Nasal operation (Surgical and medical procedures) | 1 (1)
Peripheral nerve decompression (Surgical and medical procedures) | 1 (1)
Peripheral nerve operation (Surgical and medical procedures) | 1 (1)
Plastic surgery (Surgical and medical procedures) | 1 (1)
Prosthesis implantation (Surgical and medical procedures) | 1 (1)
Salpingo-oophorectomy unilateral (Surgical and medical procedures) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 3 (3)
Shoulder operation (Surgical and medical procedures) | 4 (4)
Spinal fusion surgery (Surgical and medical procedures) | 2 (2)
Spinal operation (Surgical and medical procedures) | 3 (3)
Steroid therapy (Surgical and medical procedures) | 1 (1)
Surgery (Surgical and medical procedures) | 2 (2)
Suture insertion (Surgical and medical procedures) | 1 (1)
Tendon operation (Surgical and medical procedures) | 1 (1)
Toe operation (Surgical and medical procedures) | 2 (2)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1)
Urinary tract operation (Surgical and medical procedures) | 1 (1)
Varicose vein operation (Surgical and medical procedures) | 1 (1)
Vascular operation (Surgical and medical procedures) | 1 (1)
Vascular stent insertion (Surgical and medical procedures) | 1 (1)
Wound drainage (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 1 (1)
Angiopathy (Vascular disorders) | 3 (3)
Aortic aneurysm (Vascular disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Aortitis (Vascular disorders) | 1 (1)
Arterial disorder (Vascular disorders) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 2 (2)
Arteriosclerosis (Vascular disorders) | 5 (5)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Arteritis (Vascular disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 7 (7)
Embolism (Vascular disorders) | 1 (1)
Haemodynamic instability (Vascular disorders) | 3 (3)
Haemorrhage (Vascular disorders) | 3 (3)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 16 (17)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Hypovolaemic shock (Vascular disorders) | 2 (2)
Infarction (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 4 (4)
Ischaemia (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Pallor (Vascular disorders) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 3 (3)
Peripheral artery stenosis (Vascular disorders) | 2 (2)
Peripheral coldness (Vascular disorders) | 2 (2)
Peripheral embolism (Vascular disorders) | 1 (1)
Peripheral venous disease (Vascular disorders) | 2 (2)
Phlebitis (Vascular disorders) | 2 (2)
Shock (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 5 (5)
Vascular insufficiency (Vascular disorders) | 1 (1)
Vascular occlusion (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 4 (4)
Vasculitis necrotising (Vascular disorders) | 1 (1)
Vein disorder (Vascular disorders) | 1 (1)
Venous aneurysm (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2006-02-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT01078558/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT01078558/SAP_001.pdf